CLINICAL TRIAL: NCT06837779
Title: Clinical Evaluation of Exposed Hypersensitive Dentin Treated With Fluoride Iontophoresis Application in Comparison With Two Different Remineralizing Agents (a Randomized Clinical Trial)
Brief Title: Exposed Hypersensitive Dentin Treated With Fluoride Iontophoresis With Remineralizing Agents
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Wakwak, ASSOCITE PROFESSOR OF OPERATIVE DENTISTRY, Al-Azhar University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: FDAZUC-REC1009/2074
Record Dates: First submitted 2024-11-29; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Dentin Hypersensitivity
Keywords: hypersinsitivity; flouride iontophoresis
MeSH Terms: conditions — Dentin Sensitivity | interventions — Acidulated Phosphate Fluoride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoride Iontophoresis with Acidulated Phosphate Fluoride gel (Experimental): assessmen of iontophoresis effect on flouride ions flush to remineralization of demineralized enamel .The treatment will be assessed and recorded using VAS score immediately after the intervention, 3 months, 6 months and one year later.
  Interventions: Drug: Fluoride Iontophoresis with Acidulated Phosphate Fluoride
- remineralizing agents (Active Comparator): All remineralizing agents (Casein phosphopeptides -Amorphus Calcium Phosphate, Nano-hydroxyapatite, and Bioactive glass).
  Interventions: Drug: Remineralization with sodium fluoride varnish

INTERVENTIONS:
Drug: Fluoride Iontophoresis with Acidulated Phosphate Fluoride — Application of fluoride gel and activated with Iontophoresis electrical pole
  Arms: Fluoride Iontophoresis with Acidulated Phosphate Fluoride gel
Drug: Remineralization with sodium fluoride varnish — CASIN PHOSPHOPEPTIDE AMORPHOUS CALCIUM PHOSPHATE
  Arms: remineralizing agents

SUMMARY:
The goal of this clinical trial is to learn if the application of fluoride works to treat patients suffering from dentin hypersensitivity. It will also learn about the safety of using fluoride iontophoresis with Acidulated phosphate fluoride gel.

The main questions it aims to answer are:

Does the remineralizing agent have the ability to decrease dentin sensitivity?

Researchers will compare Fluoride Iontophoresis with Acidulated Phosphate Fluoride gel , Casein phosphopeptides-Amorphus calcium phosphate (CPP-ACP), nano-hydroxyapptite (NHAP) and -active glass in decreasing dentin hypersensitivity

.

Participants will:

* Application of remineralizing agent every 3 months
* Visit the dental clinic once every 3 months for checkups and tests

DETAILED DESCRIPTION:
Assess the efficacy of fluoride iontophoresis in remineralization in comparison with other ingredients.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 35-60 years of age.
* Each patient has 4 or more exposed roots of posterior teeth having sensitivity.
* Good oral hygiene.
* Patients who will agree to the consent and will commit to the follow-up period.
* Patients will follow instructions during study time.
* Teeth that were vital.

Exclusion Criteria:

* Patients with any systemic disease that may affect normal healing.
* Patient with bad oral hygiene, high caries index and high plaque index
* Patients participating in more than 1 dental study.
* Active carious lesions.
* Intrinsic and extrinsic stains.
* Any previous filling of selected teeth.
* Cracked and malformed teeth.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12 months
  Measurement of sensitivity was performed after each stimulus by a Visual Analogue Scale, which consists of a 10-cm long line; the minimum value is 0 and the maximum value is 10, whether the higher scores mean worse and the lower score means better outcome.
  The patient's pain limits can suffer through an external stimulus; at 0, one end represents absence of discomfort, and the other represents severe discomfort caused by certain stimuli. Each time the patient is subjected to a stimulus, he or she is requested to point at the interval from 0 to 10, a number to correspond to the pain felt. The convenience of this type of scale is to allow demonstration of the pain intensity with absolute numbers or as a percentage of a maximum value

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Wakwak, A, Principal Investigator — Alazhar Univeristy
Locations (1):
- Faculty of Dental Medicine ,Alazhar Univerisity, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
privacy of patient may be may be photo of device used in the study , photo of treatment